CLINICAL TRIAL: NCT01559636
Title: Effect of Diarrheal Disease on Bivalent Oral Polio Vaccine (bOPV) Immune Response in Infants in Nepal
Brief Title: Diarrhea and Bivalent Oral Polio Vaccine Immunity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Tribhuvan University, Nepal (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CDC-458-GID-037
Record Dates: First submitted 2012-01-04; First posted 2012-03-21 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Seroimmunity; Diarrhea; Polio
Keywords: seroconversion; oral polio vaccine; OPV; poliomyelitis; diarrhea; seroimmunity
MeSH Terms: conditions — Diarrhea; Poliomyelitis; HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diarrhea (Active Comparator): Infants with diarrhea will have blood and stool sample taken and receive zinc and ORS. They will then receive bivalent oral polio vaccine as the intervention. Four weeks later another blood sample will be drawn to measure seroconversion.
  Interventions: Biological: bivalent oral polio vaccine
- Non-diarrhea (Active Comparator): Infants without diarrhea will have blood and stool sample taken and receive multivitamins. They will then receive bivalent oral polio vaccine as the intervention. Four weeks later another blood sample will be drawn to measure seroconversion.
  Interventions: Biological: bivalent oral polio vaccine

INTERVENTIONS:
Biological: bivalent oral polio vaccine — vaccine given during immunization campaigns

SUMMARY:
Global eradication of poliomyelitis has proven to be elusive. Although 99% of cases have been eliminated since 1988, outbreaks continue to occur, and new tools are needed to accelerate eradication. One concern in this effort is that some populations have decreased immunogenicity to oral poliovirus vaccine (OPV). Past studies have shown decreased seroimmunity to trivalent OPV (tOPV) in children with diarrhea. In 2009, bivalent OPV (bOPV) was recommended for use in immunization campaigns, and will likely replace tOPV in routine immunization in 2016. However, the effect of diarrhea on seroconversion to bOPV has not been studied.

This project evaluated the effect of diarrhea on seroconversion to bOPV among infants who reside in Nepal. The investigators conducted a prospective, interventional study that assessed immune response to bOPV among infants with and without diarrhea. Immune responses were compared among infants with and without diarrhea.

This study will result in a better understanding of the factors that decrease the ability of some children to seroconvert to OPV and be protected from poliomyelitis infection.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will be including Nepali infants aged at least 6 weeks and no more than 12 months, who have received <3 doses of OPV (cumulative from routine and SIA) and present to outpatient clinics in participating study sites. Whenever possible, the child's immunization status based on the caretaker's report will be cross-checked with available immunization cards.
* Infants with diarrhea must also have:
* Current diarrhea, defined as three loose stools per day in the past 24 hours. This may include children with acute or chronic diarrhea, low grade fever, and those with intermittent vomiting who are able to tolerate oral fluids and do not present with severe dehydration on the initial visit.
* Non-diarrhea children also must:
* Present with other, non-diarrheal minor acute complaints. This can include but is not limited to children presenting for non-severe illnesses such as skin problems (e.g., rash), conjunctivitis, and mild cough, congestion, or cold. These children should be diarrhea-free for at least two weeks prior to enrolment.

Exclusion Criteria:

* Infants younger than 6 weeks or older than 12 months of age
* Infants who have received 3 or more cumulative doses of OPV (including both routine and SIAs)
* Infants who require hospitalization or are deemed too ill to participate by the study site clinician
* Infants with blood in the stool (as this may represent more severe cases including dysentery, or non-infectious severe illnesses such as intussusception)
* Infants who require IV medications for a severe illness (e.g., pneumonia); however, this does not include medications for mild or moderate illnesses, such as paracetamol, ORS, eye ointment, etc.
* Infants who have a chronic underlying illness requiring long term medications
* Infants who are unable to take any oral fluids by mouth, require IV hydration and therefore would be unable to tolerate oral medications in the study
* Infants whose caregivers do not consent, or are not present to give consent, to the study
* Infants who will not be able to return to the clinic to participate the full length of the study

Ages: 6 Weeks to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 699 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The proportion of infants who seroconvert or boost in antibody titers in the diarrhea arm compared to the non-diarrhea arm | 4 weeks after date of bOPV dose
  Seropositive: antibody titer of at least 1:8 for poliovirus type 1 or 3
  Seronegative: antibody titer of less than 1:8 for poliovirus type 1 or 3
  Seroconversion: proportion of children who change from seronegative to seropositive to types 1 or 3, four weeks after receipt of bOPV.
  Boost (increase in titer): seropositives at baseline who increase at least 4-fold in antibody titer four weeks after receipt of bOPV.

SECONDARY OUTCOMES:
Frequencies of enteric infections isolated in stool among infants with diarrhea vs. infants without diarrhea | Date of enrollment
  One stool sample will be collected from each infant the day of enrollment.
Proportion of infants seropositive after receipt of 3 doses of any oral polio vaccine | 4 weeks after date of bOPV dose
  A subset of infants who received two doses of any OPV prior to study entry, and a third dose of bOPV as part of the study, will have their seroimmunity reported. This outcome is intended as a proxy measure for seroprevalence after 3 doses of OPV, which is how the vaccine is used in routine immunization.
Proportion of infants with factors associated with poor bOPV seroconversion/boosting | 4 weeks after date of bOPV dose
  Multivariable modeling will be used to assess factors associated with poor bOPV seroconversion/boosting.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina V Cardemil, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Institute of Medicine, Kathmandu, Nepal

REFERENCES:
- [Derived] Cardemil CV, Estivariz C, Shrestha L, Sherchand JB, Sharma A, Gary HE Jr, Oberste MS, Weldon WC 3rd, Bowen MD, Vinje J, Schluter WW, Anand A, Mach O, Chu SY. The effect of diarrheal disease on bivalent oral polio vaccine (bOPV) immune response in infants in Nepal. Vaccine. 2016 May 11;34(22):2519-26. doi: 10.1016/j.vaccine.2016.03.027. Epub 2016 Apr 13. PMID 27085172
- See also: Global Polio Eradication Initiative — http://www.polioeradication.org